CLINICAL TRIAL: NCT05639751
Title: A Phase 1 Open-Label, Multi-Center, Safety and Efficacy Study of PRT3789 as Monotherapy and in Combination With Docetaxel in Participants With Advanced or Metastatic Solid Tumors With a SMARCA4 Mutation
Brief Title: PRT3789 Monotherapy and in Combo w/Docetaxel in Participants w/Advanced or Metastatic Solid Tumors w/SMARCA4 Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prelude Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT3789-01
Record Dates: First submitted 2022-11-11; First posted 2022-12-06 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Non-small Cell Lung Cancers; SMARCA4 Gene Mutation
Keywords: Advanced Solid Tumors; BRG1; BRM; Metastatic Solid Tumors; Non-Small Cell Lung Cancers; NSCLC; PRT3789; SMARCA2 Degrader; SMARCA4; Docetaxel
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRT3789 Monotherapy (Experimental): PRT3789 will be administered by intravenous infusion
  Interventions: Drug: PRT3789
- PRT3789/Docetaxel Combination (Experimental): PRT3789 and Docetaxel will be administered by intravenous infusions
  Interventions: Drug: PRT3789; Drug: Docetaxel

INTERVENTIONS:
Drug: PRT3789 — PRT3789 will be administered by intravenous infusion
Drug: Docetaxel — Docetaxel will be administered by intravenous infusion
  Arms: PRT3789/Docetaxel Combination

SUMMARY:
This is a Phase 1 dose-escalation study of PRT3789, a SMARCA2 degrader, in participants with advanced or metastatic solid tumors with loss of SMARCA4 due to truncating mutation and/or deletion. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) of PRT3789 monotherapy and in combination with docetaxel, describe any dose limiting toxicities (DLTs), define the dosing schedule, and to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) to be used in subsequent development of PRT3789.

DETAILED DESCRIPTION:
This is an open-label, multi-center, dose-escalation, first in human, Phase 1 study of PRT3789 as monotherapy and in combination with docetaxel, a SMARCA2 degrader, evaluating participants with advanced or metastatic solid tumors with loss of SMARCA4 due to truncating mutation and/or deletion. The study will evaluate escalating doses of PRT3789 until the MTD or RP2D is determined. Taking into account pharmacokinetic and pharmacodynamic data from the preceding dose levels, the dose may be escalated until a dose limiting toxicity is identified. Approximately 186 participants will be enrolled in monotherapy, dose escalation, backfill, and combination cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations (including contraception requirements), and other study procedures
* Histologically confirmed advanced, recurrent, or metastatic solid tumor malignancy with any mutation of SMARCA4 (dose escalation and combination cohorts) and loss of function mutation of SMARCA4 (backfill cohorts) by local testing that have either progress on or ineligible for standard of care therapy
* Must have measurable or non-measureable (but evaluable) disease per RECIST v1.1 for dose escalation and combination cohorts
* Must have measureable diseases per RECIST v1.1 for backfill cohort
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Willing to provide either archival or fresh tumor tissue sample
* Adequate organ function (hematology, renal, and hepatic)

Exclusion Criteria:

* Participants with solid tumors with known concomitant SMARCA2 mutation or loss of protein expression
* Clinically significant or uncontrolled cardiac disease, uncontrolled electrolyte disorders, uncontrolled or symptomatic central nervous system (CNS) metastases or leptomeningeal disease
* History of another malignancy within 3 years except for adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancies, or malignancies previously treated with curative intent and not on active therapy or expected to require treatment or recurrence during the study
* Concurrent treatment with strong or moderate CYP3A4 inhibitor or inducer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of PRT3789 monotherapy and in combination with docetaxel | Baseline through Day 21
  Dose limiting toxicities will be evaluated over the 21-day observation period
Safety and tolerability of PRT3789 monotherapy and in combination with docetaxel: AEs, CTCAE Assessments | Baseline through approximately 3 years
  Safety and tolerability will be evaluated by incidence of DLTs, laboratory measurements, dose interruption, modification, and discontinuation due to adverse events (AEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Maximum tolerated dose (MTD)/ Recommended phase 2 dose (RP2D) of PRT3789 monotherapy and in combination with docetaxel | Baseline through approximately 3 years
  The MTD/RP2D will be established for further investigation in participants with advanced solid tumors

SECONDARY OUTCOMES:
Efficacy of PRT3789 monotherapy and in combination with docetaxel: Objective response rate (ORR) | Baseline through approximately 3 years
  Best overall response of either complete response (CR) or partial response (PR), as assessed by the investigator per RECIST v1.1
Efficacy of PRT3789 monotherapy and in combination with docetaxel: Progression-free survival (PFS) | Baseline through approximately 3 years
  Duration from Day 1 to the earliest date of first disease progression, as assessed by the investigator per RECIST v1.1, discontinuation because of disease progression, or death due to any cause
Efficacy of PRT3789 monotherapy and in combination with docetaxel: Clinical benefit rate (CBR) | Baseline through approximately 3 years
  Best overall response of CR, PR, or durable stable disease (24 weeks or longer duration), as assessed by the investigator per RECIST v1.1
Efficacy of PRT3789 monotherapy and in combination with docetaxel: Duration of response (DOR) | Baseline through approximately 3 years
  Duration from time of first observed response (CR or PR) to the earliest date of disease progression, as assessed by the investigator per RECIST v1.1, or death due to any cause
Pharmacokinetic profile of PRT3789 monotherapy and in combination with docetaxel: Maximum observed plasma concentration | Baseline through approximately 3 years
  Pharmacokinetics will be calculated including the maximum observed plasma concentration
Pharmacokinetic profile of PRT3789 monotherapy and in combination with docetaxel: Area under the curve | Baseline through approximately 3 years
  Pharmacokinetics will be calculated including the area under the plasma concentration versus time curve (AUC)
Pharmacodynamic effect of PRT3789 monotherapy and in combination with docetaxel: Target engagement | Baseline through approximately 3 years
  Pharmacodynamic effect of PRT3789 monotherapy and in combination with docetaxel demonstrating target engagement by assessment of SMARCA2 protein in peripheral blood mononuclear cells (PBMCs) and tumor tissue

CONTACTS AND LOCATIONS:
Locations (32):
- United States (20):
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - AdventHealth Medical Group Oncology Research at Celebration, Celebration, Florida
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - New York Presbyterian Hospital - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia
- France (5):
  - lnstitut Bergonie Centre Regionale de Lutte Contre le cancer, Service Oncologie-Medicale, Bordeaux
  - Centre Leon Berard, Lyon
  - lnstitut Paoli Calmettes, Marseille
  - Oncopole Claudius Regaud IUCT ONCOPOLE, Toulouse
  - Institut Gustave Roussy, Villejuif
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - National Cancer Centre Singapore, Singapore, Singapore
- Spain (4):
  - START Barcelona - HM Nou Delfos, Barcelona, Barcelona
  - START MADRID - FJD Hospital Universitario Fundacion Jimenez Diaz, Madrid, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid, Madrid
  - Hospital Universitario Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No